CLINICAL TRIAL: NCT03572426
Title: Ion Channel Genetic Biomarkers: Diagnostic Capabilities in the Assessment of Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Sigma Theta Tau (Unknown)
Responsible Party: Sponsor
Other Study IDs: 17-1578
Record Dates: First submitted 2018-06-13; First posted 2018-06-28 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Buccal Swab collect with genotyping done by SNaPshot.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bipolar: Diagnosed as having at least 1 lifetime manic episode by the MINI
  Interventions: Other: genotyping all subjects
- Depression: Diagnosed as having at least 1 Major Depressive Episode by the MINI
  Interventions: Other: genotyping all subjects
- Healthy Controls: Does not meet Criteria for any mood disorder diagnosis (MDD, BD, dysthymia)
  Interventions: Other: genotyping all subjects

INTERVENTIONS:
Other: genotyping all subjects — genotyping using SNaPshot genotyping method.

SUMMARY:
Genotype 164 adults to evaluate six selected single nucleotide polymorphisms (SNPs) (rs1006737, rs10994336, rs10994133, rs2238071, rs1051375, rs1024582) for use as a genetic biomarker to differentiate between bipolar depression and unipolar depression.

DETAILED DESCRIPTION:
Adults ages 18-80 will be recruited if they are diagnosed with bipolar disorder, major depression, or have no mood symptoms. The adults will undergo a diagnostic interview, the Mini International Neuropsychiatric Interview (MINI) for the diagnosis. The subjects will also complete the Adverse Childhood Events Scale to evaluate for a genetic x environmental interaction in detecting bipolar disorder at initial assessment. Genotyping will be done by SNaPshot genotyping method and genetic sample will be collected via buccal swab.

ELIGIBILITY:
Inclusion Criteria:

* presenting to one of 4 Denver Metro Area clinics
* Subjects must fall into one of 3 diagnostic categories, bipolar, MDD, or no mood symptoms.

Exclusion Criteria:

* Inability to provide informed consent
* history of TBI
* history of untreated seizure disorder
* substance abuse in the last 8 hours
* moderate-severe substance abuse disorder diagnosed in the last 6 months

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Caucasian and Latino
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Logistic Regression | 1 year
  Logistic regression will be used to examine a genetic risk score using a risk allele count as the independent variable, with a diagnosis of BD versus MDD versus those with no mood diagnosis as the dependent variable.

SECONDARY OUTCOMES:
Genetic Risk Score | 1 year
  Genetic risk score of selected SNPsrs1006737, rs10994336, rs10994133, rs2238071, rs1051375, rs1024582
Family History | 1 year
  Positive family history of bipolar disorder in a first degree relative
Adverse Childhood Experiences Scale | 1 year
  0-10 item scale assessing for adversity experienced during childhood

CONTACTS AND LOCATIONS:
Overall Officials: Kristiana Avery, PhD-c, Principal Investigator — University of Colorado, Denver
Locations (1):
- Helen and Arthur E Johnson Depression Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided